CLINICAL TRIAL: NCT05826522
Title: Preliminary Monocentric Study for the Validation of the Circuit of Examinations and Analyzes of Samples in Perspective of Large-scale Application for Better Classification of Airway Diseases
Brief Title: Study for the Validation of the Circuit of Examinations and Analyzes for Better Classification of Airway Diseases
Acronym: BABY-ROAD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hopital Foch (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-A01154-39
Record Dates: First submitted 2023-02-08; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Airway Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, faces ,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- asthmatics and asthmatics previously
  Interventions: Other: observationnal
- COPD (chronic obstructive pulmonary disease) patients
  Interventions: Other: observationnal
- cystic fibrosis patients
  Interventions: Other: observationnal
- patients with immunodeficiency with bronchial obstruction
  Interventions: Other: observationnal
- lung transplant recipients with obstructive chronic lung allograft rejection (O-CLAD)
  Interventions: Other: observationnal

INTERVENTIONS:
Other: observationnal — cohort of blood collection and severals exams

SUMMARY:
ADs (airway diseases) are a group of progressive diseases that lead to a decline of lung function, accelerated by recurrent exacerbations, which can lead to death. ADs include a number of different conditions including asthma, chronic obstructive pulmonary disease (COPD), cystic fibrosis (CF), bronchiectasis and bronchiolitis frequently related to immune difciency or hematopoietic stem cell transplantations (HSCT), and obstructive chronic lung allograft dysfunction (O-CLAD). The financial burden of ADs is monumental. It is imperative to prevent exacerbations and decline in lung function to reduce ADs mortality and morbidity. The vast amount of knowledge accumulated over the last several years in both biotechnology and digital intelligence, has afforded the evidence of the presence of various treatable traits spread among ADs, that imposes to reassess ADs. BABY-ROAD study proposes to take advantage of these advances to test the feasibility of sampling and exploring ADs patients with multisource data. Baby-ROAD study will be preliminary to the ROAD study that will propose to reclassify ADs into new clusters pertinent for preventive, personalized and participative care.

DETAILED DESCRIPTION:
Study population: Patients who are part of the group of ADs. This group of progressive diseases lead to a decline of lung function which is accelerated by recurrent exacerbations, which can in turn lead to death. The study population will include severe asthmatics and asthmatics previously hospitalized at least once in 2016 - 2019, COPD (chronic obstructive pulmonary disease) patients previously hospitalized at least once in 2016 - 2019, cystic fibrosis patients, patients with immunodeficiency with bronchial obstruction, lung transplant recipients with obstructive chronic lung allograft rejection (O-CLAD) and hematopoietic stem cell transplant recipients with bronchial obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Severe asthmatics + asthmatics previously hospitalized at least once in 2016 - 2019
* COPD patients previously hospitalized at least once in 2016 - 2019 Cystic fibrosis patients, patients with immunodeficiency, without bone marrow transplantation, and with AD determined upon bronchial obstruction (FEV1/FVC < 70%).
* Lung transplant recipients with obstructive chronic lung allograft rejection (O-CLAD)
* Hematopoietic stem cell transplant recipients with AD determined upon bronchial obstruction.
* Patients already followed-up in pulmonology clinic at the Foch Hospital
* Patients understanding the French language
* Patients having signed an informed consent form prior to any study specific procedure
* Patients being covered by a national health insurance

Exclusion Criteria:

* COPD patients previously hospitalized but before 2016
* Immunocompromised patients, having had a bone marrow transplant and suffering from AD determined by bronchial obstruction (FEV1/FVC > 70%).
* Patients weighing less than 50 kg
* Pregnant women
* Patients who are not followed in pulmonology consultation at Foch Hospital
* Patients don't understanding the French language
* Don't being covered by a national health insurance
* Being deprived of liberty or under guardianship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are part of the group of ADs. This group of progressive diseases lead to a decline of lung function which is accelerated by recurrent exacerbations, which can in turn lead to death. The study population will include severe asthmatics and asthmatics previously hospitalized at least once in 2016 - 2019, COPD (chronic obstructive pulmonary disease) patients previously hospitalized at least once in 2016 - 2019, cystic fibrosis patients, patients with immunodeficiency with bronchial obstruction, lung transplant recipients with obstructive chronic lung allograft rejection (O-CLAD) and hematopoietic stem cell transplant recipients with bronchial obstruction
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
To validate the circuit of examinations and sample analysis within the Foch hospital to show that this study is feasible on a large scale (600 patients) | one year
  ensure that all patients included have undergone the examinations indicated in the protocol

SECONDARY OUTCOMES:
To show that the small number of patients (50) partly achieves the objectives of the next "ROAD 2028" multicentric trial (600 patients) | one year
  ensure that all patients included have undergone the examinations indicated in the protocol